CLINICAL TRIAL: NCT01251081
Title: Effect of the Intensity of Continuous Renal Replacement Therapy in Patients With Sepsis and Acute Kidney Injury: Single-center Randomized Clinical Trial
Brief Title: Effect of the Intensity of Continuous Renal Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhejiang University (Other)
Purpose: Treatment
Other Study IDs: VHVHF
Record Dates: First submitted 2010-11-30; First posted 2010-12-01 (Estimated); Last update posted 2010-12-01 (Estimated); Status verified 2004-01

CONDITIONS: Optimal Intensity of Renal Replacement Therapy on Sepsis Patients
Keywords: high volume hemofiltration; sepsis; acute kidney injury; survival
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- extra high volume hemofiltration (Experimental): extra high volume hemofiltration (85 mL/kg/h, EHVHF)
  Interventions: Other: extra high volume hemofiltration
- high volume hemofiltration (Sham Comparator): high volume hemofiltration (50 mL/kg/h, HVHF)
  Interventions: Other: high volume hemofiltration

INTERVENTIONS:
Other: extra high volume hemofiltration — extra high volume hemofiltration (85 mL/kg/h, EHVHF)
  Arms: extra high volume hemofiltration
Other: high volume hemofiltration — high volume hemofiltration (50 mL/kg/h, HVHF)
  Arms: high volume hemofiltration

SUMMARY:
In patients with sepsis and AKI, increasing the intensity of renal replacement therapy from 50 mL/kg/h (HVHF) to 85 mL/kg/h (EHVHF)will increase the survival at 28 days and 90 days.

ELIGIBILITY:
Inclusion Criteria:

met at least one of the following criteria: oliguria (urine output less than 100 mL in a 6 h period and unresponsive to fluid resuscitation), serum potassium concentration more than 6.5 mmol/L, severe acidemia (pH < 7.2), serum creatinine more than 250 µmol/L, or presence of severe organ edema (e.g. pulmonary edema).

Exclusion Criteria:

* were presence of a malignant tumor, chronic renal insufficiency (serum creatinine >133 µmol/L), or receiving any kind of renal replacement therapy before randomization.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2004-01; Primary Completion 2009-08 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
90 days survival
  The primary study outcome was death from any cause within 90 days. Results were analyzed by Kaplan-Meier survival curves

SECONDARY OUTCOMES:
length of stay in the ICU and hospital
  Secondary outcomes were length of stay in the ICU and hospital and renal outcome of survivors at 90 days after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: jianghua chen, MD, Study Director — Kidney disease center, the first affiliated hospital, medical college of Zhejiang university
Locations (1):
- Kidney disease center, the first affiliated hospital, medical college of Zhejiang university, Hangzhou, Zhejiang, China